CLINICAL TRIAL: NCT06263699
Title: Comparing the Accuracy of Clinical Goniometry and Goniometric Measurement on Standardised Images in Dupuytren's Disease
Brief Title: Goniometry and Goniometric Measurement on Standardised Images in Dupuytren's Disease
Acronym: Goniometry
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S68225
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Dupuytren's Disease
MeSH Terms: conditions — Dupuytren Contracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with diagnosed Dupuytren's disease: Range of motion measurement of the MCP and PIP joints in digits 4 and 5
  Interventions: Procedure: ROM measurement of the MCP and PIP joints in digits 4 and 5

INTERVENTIONS:
Procedure: ROM measurement of the MCP and PIP joints in digits 4 and 5 — standardised picture of the hand in maximal active extension, with the back of the hand positioned on the table's surface
  Other Names: Standardised picture of the hand

SUMMARY:
Measuring range of motion (ROM) is essential in detecting musculoskeletal deficits, monitoring the effects of treatment and progression of the disease. In Dupuytren's disease the active and passive extension deficits (AED, PED) of digits 4 and 5 are usually clinically measured using a universal, short arm goniometer which is considered the standard of care. Using the goniometer can be time consuming. Measuring the extension deficit on a standardised picture could improve follow up, since it is a faster and easier process to take a picture and upload it to the patients files. Though this gives rise to the question whether this kind of measurement would be equally accurate and reliable in comparison to regular clinical measurement using a goniometer.

DETAILED DESCRIPTION:
Measuring range of motion (ROM) is essential in detecting musculoskeletal deficits, monitoring the effects of treatment and progression of the disease. In Dupuytren's disease the active and passive extension deficits (AED, PED) of digits 4 and 5 are usually clinically measured using a universal, short arm goniometer which is considered the standard of care. Using the goniometer to measure the extension deficit of both fingers, for both the proximal interphalangeal (PIP) and metacarpophalangeal (MCP) joint can be a time consuming process. A lot of clinicians have limited time per patient, which leads to partially or completely missing data due to not performing the measurements. Measuring the extension deficit on a standardised picture could improve follow up, since it is a faster and easier process to take a picture and upload it to the patients files. Though this gives rise to the question whether this kind of measurement would be equally accurate and reliable in comparison to regular clinical measurement using a goniometer. Establishing the difference between both methods is essential to monitor change, which makes a statistical comparison of accuracy of both methods very valuable for patients with Dupuytren's disease. Furthermore, a lot of clinicians have collected and stored standardised pictures of their patient's hands over the years. Therefore this study could solidify the available data through these images, which provide valuable information for future follow up. Furthermore, proper patient education could provide the clinician with standardised images taken by the patient himself, leading to improved follow up, if images and clinical measurement prove to be equally accurate.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age
* Current AED in digit 4 or 5, in the MCP or PIP joint

Exclusion Criteria:

* Abnormalities to the fingers other than Dupuytren's disease which make goniometry impossible (e.g. amputation, arthrodesis of finger joints, deformations due to rheumatoid arthritis etc.)
* Patient's unable to give a written participating consent.
* Younger than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed Dupuytren's disease
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Active Extension Deficits (AED) | Baseline
  AED in the MCP and PIP joints of digit 4 and 5 are measured by using a goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Ilse Degreef, Prof. Dr, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitaire Ziekenhuizen KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No